CLINICAL TRIAL: NCT04361461
Title: Hydroxychloroquine or Hydroxychloroquine Associated With Azithromycin for Inpatients With Moderate or Severe Lung Disease Due to SARS-CoV-2 (COVID-19)
Brief Title: Use of Hydroxychloroquine Alone or Associated for Inpatients With SARS-CoV2 Virus (COVID-19)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: This study was canceled before enrollment due to a decision by the Sponsor
Sponsor: Apsen Farmaceutica S.A. (Industry)
Collaborators: Federal University of São Paulo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APS000/2020
Record Dates: First submitted 2020-04-22; First posted 2020-04-24 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-06

CONDITIONS: Coronavirus Infections; SARS-CoV 2; SARS (Severe Acute Respiratory Syndrome); Pulmonary Disease
MeSH Terms: conditions — Coronavirus Infections; Severe Acute Respiratory Syndrome; Lung Diseases | interventions — Hydroxychloroquine; Azithromycin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Hydroxychloroquine (400 mg)
  Interventions: Drug: Hydroxychloroquine Sulfate
- Group 2 (Experimental): Hydroxychloroquine (400 mg) + azithromycin (500 mg)
  Interventions: Drug: Hydroxychloroquine Sulfate + Azythromycin

INTERVENTIONS:
Drug: Hydroxychloroquine Sulfate — 400 mg orally, every 12 hours x 2 doses (loading dose) and then 400 mg, once daily, orally, for 10 days.
  Other Names: Reuquinol®
  Arms: Group 1
Drug: Hydroxychloroquine Sulfate + Azythromycin — 400 mg, orally, every 12 hours x 2 doses (loading dose) and then 400 mg, once a day, orally, for 10 days associated with azithromycin, intravenously or orally, 500 mg / day, for 1 day and then 250mg / day for another 4 days.
  Other Names: Reuquinol® + Azythromycin
  Arms: Group 2

SUMMARY:
The Severe Acute Respiratory Syndrome CoronaVirus 2 (SARS-CoV2) has been identified in Wuhan, China, which causes severe pulmonary complications and flu syndrome, which has spread rapidly to all continents. Approximately 25% of hospitalized patients require treatment in intensive care units and 10% require mechanical ventilation. The diagnosis is made by the molecular polymerase chain reaction test. However, diagnostic tests are limited. The clinical care of the patient with COVID-19 is similar to that of patients with severe infectious respiratory complications, consisting of support and oxygen supplementation. Several medications have been tested as remdesivir, a pro-drug nucleoside, which acts by inhibiting viral RNA transcription, although a recently published study has shown no benefit. China recently approved the use of favipiravir, an antiviral used for influenza, as an experimental therapy for COVID-19. Hydroxychloroquine is a drug with great potential treatment, as it can inhibit the pH-dependent steps of replication of various viruses, with a potent effect on SARS-CoV infection and spread. In this way, the present study will evaluate the safety and efficacy of the hydroxychloroquine in patients with symptomatic SARS-Cov2.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged > 18 years;
* Patients with flu syndrome (fever greater than 37.8C or feverish feeling referred by the patient associated with at least 1 respiratory symptom: cough, difficulty breathing, sputum production, nasal or conjunctival congestion, difficulty swallowing, sore throat, runny nose, signs cyanosis, flapping of the nose and dyspnoea);
* Diagnosis confirmed by real-time PCR or suspected COVID-19;
* Hospitalized patients with:
* Moderate disease: hypoxemia with O2 saturation <93% in room air and / or respiratory rate greater than or equal to 24 incursions per minute and / or radiological evidence of pneumonia with pulmonary impairment less than 50%;

or

* Serious illness: Hospitalized patients with hypoxemia with O2 saturation <93% in room air and / or respiratory rate greater than or equal to 24 incursions per minute with radiological evidence of pneumonia with pulmonary involvement above 50% and / or the presence of sepsis ( organ failure) or need for invasive mechanical ventilation.

Exclusion Criteria:

* Mild cases of flu-like syndrome that do not require hospitalization or O2 saturation greater than or equal to 93% and without radiological evidence of pneumonia;
* Liver failure or elevation of transaminases greater than 5 times;
* Cardiac patients with electrocardiogram with extended QT interval;
* Pregnant women;
* Use in the last 30 days of hydroxychloroquine or azithromycin;
* Allergy to hydroxychloroquine or azithromycin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04-30 (Estimated); Primary Completion 2020-11-04 (Estimated); Study Completion 2020-11-04 (Estimated)

PRIMARY OUTCOMES:
Individual response rate | 14 days after randomization
  The individual response rate regarding the World Health Organization Ordinal Scale assessment from basal to 14th Day.

SECONDARY OUTCOMES:
All-cause mortality | 28 days after randomization
  All-cause mortality rates at Day 28th after randomization
Duration of mechanical ventilation | baseline
  Number of days that the patient was on mechanical ventilation which was under ventilation from basal line
Proportion of patients which needed mechanical ventilation during study | hospitalization within 28 days
  Proportion of patients who do not receive mechanical ventilation at the beginning of the study and then needed mechanical ventilation during hospitalization.
World Health Organization (WHO) Ordinal scale | 28 days after inclusion and compared to baseline
  The ordinal scale is an assessment of the clinical status at the first clinical evaluation in a clinical study. The scale is as follows: 1) Death; 2) Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); 3) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 4) Hospitalized, requiring supplemental oxygen; 5) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 6) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 7) Not hospitalized, limitation on activities and/or requiring home oxygen; 8) Not hospitalized, no limitations on activities.
Duration of hospitalization | hospitalization within 28 days
  Length of hospital stay in days for hospitalization
Rates of drug discontinuation | hospitalization within 28 days
  Rates of drug discontinuation in all causes under study

OTHER OUTCOMES:
Rates of serious adverse events | Day 14th
  Rates of serious adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Apsen Farmacêutica S.A., São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No